CLINICAL TRIAL: NCT03562676
Title: VESTIBULAR EVOKED MYOGENIC POTENTIALS IN ALTERED GRAVITY
Acronym: VEMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-161
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- weightlessness (Experimental)
  Interventions: Other: weightlessness

INTERVENTIONS:
Other: weightlessness — parabolic flight

SUMMARY:
Recently, new clinical testing of saccular and utricular function have been developed and validated, the so-called vestibular-evoked myogenic potentials - VEMP (Brantberg et al. 2009, Cornell et al. 2009, Curthoys 2010, Manzari et al. 2012). Among them, the cervical VEMP (cVEMP) are short-latency electromyographic (EMG) modulations of the contracted sternocleidomastoid muscles in responses to vibration applied on the forehead. The clinical literature suggests that cVEMP are almost entirely saccular in origin (Halmagyi et al 1995).

The aim of our research is to evaluate changes in the otolith function in microgravity and hypergravity using this clinical test. Cervical vestibular-evoked myogenic potentials (cVEMP) will be recorded by surface EMG electrodes in response to bone conducted vibration to specifically assess saccular function (Halmagyi et al 1995). The primary measures will include muscle activity response amplitudes and the stimulus intensity threshold at which the cVEMP is detected.

Given that there is an off-loading of the saccules in microgravity and an increased loading in hypergravity, we hypothesize that there will be a reduction in cVEMP amplitude in microgravity and an increase in cVEMP amplitude in hypregravity compared to normal gravity. These changes in amplitude will be accompanied by changes in the threshold of the stimulus level required to elicit a cVEMP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 67
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* With normal cVEMP
* Who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women (urine pregnancy test for women of childbearing potential)

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
vestibular-evoked myogenic potentials (P13-N23) | baseline
  amplitude and treshold

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No